CLINICAL TRIAL: NCT03139318
Title: Phase I Clinical Trial of GRID Therapy in Pediatric Osteosarcoma of the Extremity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 and the resulting administrative issues, it is not feasible to continue the study.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 205993
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Osteosarcoma in Children; Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- GRID Radiotherapy (Experimental): Patients will be treated with GRID Radiotherapy
  Interventions: Radiation: GRID radiotherapy

INTERVENTIONS:
Radiation: GRID radiotherapy — Patients will be treated with GRID radiotherapy

SUMMARY:
The primary objective of this study is to evaluate the toxicity profile of GRID therapy using dose levels of 10Gy, 15 Gy and 20Gy in pediatric osteosarcoma of the extremity.

DETAILED DESCRIPTION:
Subjects will receive GRID radiotherapy. GRID radiation therapy is considered a standard radiation therapy method however is not typically used in pediatric osteosarcoma patients. This protocol will evaluate whether or not the use of this therapy will provide benefit to this patient population.

ELIGIBILITY:
Inclusion Criteria:

* History of cytological or histological documentation of non-metastatic extremity osteosarcoma.
* 5-21 years of age.
* Subject is eligible for routine chemotherapy and routine surgery for the treatment of non-metastatic extremity osteosarcoma
* Informed consent is obtained

Exclusion Criteria:

* Females with a positive urine pregnancy test.
* Unable to comply with study procedures

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Harrell, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRID Radiotherapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GRID Radiotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicities Associated With GRID Radiotherapy
Description: The study endpoint is dose-limiting toxicity (DLT), which is defined as a treatment-related AE of Grade 3 or higher.
Time Frame: An average of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | GRID Radiotherapy
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 90 days (+/- 7 days) post surgery
Description: The PI must be notified within 24 hours of learning of any serious adverse events, regardless of attribution, occurring during the study. The IRB must be notified within 10 business days of any unanticipated problems involving risk to subjects or others. All other adverse events, such as those that are expected, or are unlikely or definitely not related to the study participation, are to be reported annually as part of regular IRB continuing review.
Arm/Group | GRID Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRID Radiotherapy (N=1)
Surgical wound breakdown (Grade 2) (Surgical and medical procedures) | 1 (1)
Surgical wound breakdown (Grade 3) (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT03139318/Prot_SAP_ICF_000.pdf